CLINICAL TRIAL: NCT05021198
Title: Epidemiology, Clinical and Radiological Presentation and Long-term Prognosis of Cerebral Venous Thrombosis in a Norwegian Population (NoCVT)
Brief Title: The Norwegian Cerebral Venous Thrombosis Study
Acronym: NoCVT
Status: Recruiting | Type: Observational
Sponsor: University Hospital, Akershus (Other)
Collaborators: Oslo University Hospital (Other); Haukeland University Hospital (Other); Drammen sykehus (Other); Sorlandet Hospital HF (Other Government); St. Olavs Hospital (Other); Nordlandssykehuset HF (Other); University Hospital of North Norway (Other); University of Oslo (Other); Rigshospitalet, Denmark (Other); Hospital de Santa Maria, Portugal (Other); Sykehuset Innlandet HF (Other); Molde Hospital (Other); Helse Stavanger HF (Other Government); Sykehuset Telemark (Other Government); Sykehuset i Vestfold HF (Other)
Responsible Party: Principal Investigator, Espen Saxhaug Kristoffersen, Principle Investigator, University Hospital, Akershus
Other Study IDs: NoCVT
Record Dates: First submitted 2021-05-27; First posted 2021-08-25 (Actual); Last update posted 2025-02-05 (Actual); Status verified 2025-02

CONDITIONS: Cerebral Vein Thrombosis; Cerebral Venous Sinus Thrombosis
MeSH Terms: conditions — Intracranial Thrombosis

STUDY DESIGN:
Observational Model: Cohort | Time Perspective: Other
Oversight: Data Monitoring Committee: No | FDA-regulated Drug: No | FDA-regulated Device: No | US Export: No

SUMMARY:
The NoCVT study will investigate CVT (2014-2023) in a large Norwegian population (> 3 millions) using several approaches combining existing health registries, clinical databases and new prospectively collected clinical data to explore epidemiology, risk factors, diagnostics, treatment, and the long-term prognosis of CVT.

DETAILED DESCRIPTION:
A retrospective hospital-based chart review will be conducted at 13 different hospitals covering all four health regions and more than 3 million inhabitants in Norway. These 13 hospitals are Akershus University Hospital, Haukeland University Hospital. Oslo University Hospital (Ullevål), Sørlandet Hospital Kristiansand, Drammen Hospital, St.Olavs Hospital, Nordlandsykehuset Bodø, University Hospital of North Norway, Innlandet Hospital Lillehammer, Tønsberg Hospital, Telemark Hospital (Skien), Molde Hospital and Stavanger University Hospital.

A search will be made in the clinical database for patients with the relevant diagnosis of CVT in the period between January 1, 2014, and December 31, 2023. Data from hospital charts will be linked with data from Statistics Norway (SSB), FD-Trygd, and Norwegian Prescription Database (NorPD). Using this combination of clinical data and health registries will make it possible to describe risk factors, clinical and radiological presentation, treatment and short-term outcome in a large Norwegian CVT cohort.

Further, data from hospitals will be linked with data from SSB, FD-Trygd, NorPD, Norwegian Patient Registry (NPR) and Cause of Death Registry (DÅR) up to five years after CVT. Using this methodology will make it possible to investigate overall long-term prognosis and outcomes in terms of mortality, health care utilisation, medication use and working situation up to five years after CVT in a large Norwegian cohort.

Lastly, a prospective follow-up study will include patients that have been diagnosed with CVT at the NoCVT hospitals during 2019-2023. By combining the collected data from the retrospective hospital chart review with the new follow-up interviews and self-reported questionnaires it will be possible to describe quality of life, vocational outcomes, psychological distress, depression, insomnia and disease-related disability in CVT.

ELIGIBILITY:
Inclusion Criteria:

* A diagnosis of CVT 2014-2023 from the 13 participating primary hospitals

Exclusion Criteria:

* none

Sex: All | Healthy Volunteers: No
Age Groups: Child, Adult, Older Adult
Study Population: A retrospective hospital-based chart review will be conducted at 13 different hospitals covering approximately 3 million inhabitants in Norway.
  More precis, a validated ICD-10 search will be made in the clinical database for patients with the diagnosis of CVT in the period between January 1, 2014, and December 31, 2023. Data from the clinical databases at these hospitals will be linked with the mandatory National Health Registries for baseline data and prospectively collected follow-up data. The National Health Registries involved are Statistics Norway (SSB), Norwegian Prescription Database (NorPD), Norwegian Patient Registry (NPR) and Cause of Death Registry (DÅR).
  In addition a clinical follow-up interview will be conducted with emphasis on long-term outcomes.
Sampling Method: Probability Sample
Enrollment: 600 (Estimated)
Dates: Start 2014-01-01 (Actual); Primary Completion 2026-12-31 (Estimated); Study Completion 2027-01 (Estimated)

PRIMARY OUTCOMES:
Mortality of CVT in a Norwegian population | Baseline, 3 months, 12 months, 24 months and 5 years
  Number dead vs total number of cases

SECONDARY OUTCOMES:
Health care utilisation after CVT | Baseline to five years
  Number of new health care system contacts among CVT cases
Re-admission after CVT | Baseline to five years
  Number of new re-admission among CVT cases
New diagnosis after CVT | Baseline to five years
  Type of new diagnosis among CVT cases
New prescriptions after CVT | Baseline to five years
  Type of new prescriptions among CVT cases
Nursing home after CVT | Baseline to five years
  Number of CVT cases in need for nursing home
Use of anti-coagulation in the long-term after CVT | Baseline to five years
  Number of cases with CVT using anti-coagulation
Use of anti-platelet therapy in the long-term after CVT | Baseline to five years
  Number of cases with CVT using anti-platelet therapy
Use of painkillers in the long-term after CVT | Baseline to five years
  Number of cases with CVT using painkillers
Use of headache prophylactics in the long-term after CVT | Baseline to five years
  Number of cases with CVT using headache prophylactics
Use of anti-epileptic drugs in the long-term after CVT | Baseline to five years
  Number of cases with CVT using anti-epileptic drugs
Use of anti-depressants in the long-term after CVT | Baseline to five years
  Number of cases with CVT using anti-epileptic drugs
Sick-leave after CVT | Baseline to five years
  Number of cases with CVT on sick-leave
Disability pension after CVT | Baseline to five years
  Number of cases with CVT on disability pension
Headache after CVT | Baseline to five years
  Type and frequency
Headache-related quality of life after CVT | Baseline to five years
  Migraine Disability Assessment Score and Headache Impact Test-6
Seizure/epilepsy after CVT | Baseline to five years
  Type and frequency
Epilepsy-related quality of life after CVT | Baseline to five years
  Quality of Life in Epilepsy Inventory-31
Quality of life after CVT | Baseline to five years
  EuroQoL 5
Psychological distress after CVT | Baseline to five years
  Patient Health Questionnaire-9 and Hospital Anxiety and Depression Scale
Sleep problems after CVT | Baseline to five years
  Bergen Insomnia Scale

CONTACTS AND LOCATIONS:
Overall Officials: Espen Saxhaug Kristoffersen, MD, PhD, Principal Investigator — University Hospital, Akershus
Locations (1):
- Akershus University Hospital, Lørenskog, Norway

IPD SHARING:
Plan to Share IPD: Undecided

REFERENCES:
- [Background] Kristoffersen ES, Harper CE, Vetvik KG, Zarnovicky S, Hansen JM, Faiz KW. Incidence and Mortality of Cerebral Venous Thrombosis in a Norwegian Population. Stroke. 2020 Oct;51(10):3023-3029. doi: 10.1161/STROKEAHA.120.030800. Epub 2020 Sep 4. PMID 32883194